CLINICAL TRIAL: NCT06112613
Title: Improving Medication Adherence in Metastatic Breast Cancer Using a Connected Customized Treatment Platform (CONCURxP)
Brief Title: Mobile Health for Adherence in Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EAQ221CD; NCI-2023-02646 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAQ221CD (Other: ECOG-ACRIN Cancer Research Group); ECOG-ACRIN-EAQ221CD (Other: DCP); EAQ221CD (Other: CTEP); R01CA262312 (NIH); UG1CA189828 (NIH)
Record Dates: First submitted 2023-10-10; First posted 2023-11-01 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Breast Carcinoma; HER2-Negative Breast Carcinoma; Hormone Receptor-Positive Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Health Promotion; Educational Status; Interviews as Topic; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARM A (Enhanced usual care) (Experimental): Patients use the WiseBag medication dispenser and receive access to educational materials every 4 weeks over 12 months.
  Interventions: Other: Electronic Health Record Review; Other: Health Promotion and Education; Procedure: Health Telemonitoring; Other: Survey Administration
- ARM B (CONCURxP program) (Experimental): Patients use the WiseBag medication dispenser and receive personalized text message reminders, medication tracking and healthcare provider follow ups as part of the CONCURxP platform over 12 months. Patients may complete an interview over 20-30 minutes within 6 months of study completion.
  Interventions: Other: Electronic Health Record Review; Procedure: Health Telemonitoring; Other: Interview; Behavioral: Patient Navigation; Other: Survey Administration; Other: Text Message-Based Navigation Intervention
- ARM C (Non-patient interview) (Experimental): Participants complete an interview over 20-30 minutes 15-39 months post-first patient enrollment.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Electronic Health Record Review — Ancillary studies
  Arms: ARM A (Enhanced usual care); ARM B (CONCURxP program)
Other: Health Promotion and Education — Receive access to educational materials
  Arms: ARM A (Enhanced usual care)
Procedure: Health Telemonitoring — Utilize the WiseBag medication dispenser
  Arms: ARM A (Enhanced usual care); ARM B (CONCURxP program)
Other: Interview — Complete an interview
  Arms: ARM B (CONCURxP program); ARM C (Non-patient interview)
Behavioral: Patient Navigation — Receive healthcare provider follow ups as part of the CONCURxP program
  Other Names: Patient Navigator Program
  Arms: ARM B (CONCURxP program)
Other: Survey Administration — Ancillary studies
  Arms: ARM A (Enhanced usual care); ARM B (CONCURxP program)
Other: Text Message-Based Navigation Intervention — Receive personalized text message reminders related to their medication tracking as part of the CONCURxP program
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation
  Arms: ARM B (CONCURxP program)

SUMMARY:
This clinical trial compares the use of the connected customized treatment platform (CONCURxP), consisting of using a medication monitoring device called WiseBag along with text message reminders for missed or extra medication events, to enhanced usual care (EUC), where patients only use the WiseBag, to monitor medication adherence in patients with metastatic breast cancer who are taking a CKD4/6 inhibitor. To ensure CDK4/6 inhibitors achieve their full clinical benefit, patients need to take them as prescribed, following a complex treatment schedule. Forgetfulness was the most common reason reported for medication non adherence. Using the WiseBag along with CONCURxP or enhanced usual care may improve medication adherence in patients with metastatic breast cancer who are taking a CKD4/6 inhibitor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare CDK4/6 inhibitors (CDK4/6i) adherence at 12 months after completion of the baseline survey captured using electronic monitoring between the EUC (Arm A) and CONCURxP (Arm B) arms.

SECONDARY OBJECTIVES:

I. To compare CDK4/6i adherence at 12 months after completion of the baseline survey captured through self-report between the EUC (Arm A) and CONCURxP (Arm B) arms.

II. To compare CDK4/6i persistence at 12 months after completion of the baseline survey captured using electronic monitoring between the EUC (Arm A) and CONCURxP (Arm B) arms.

III. To compare symptom burden at 12 months between the EUC (Arm A) and CONCURxP (Arm B) arms.

IV. To compare quality of life at 12 months between the EUC (Arm A) and CONCURxP (Arm B) arms.

V. To compare patient-provider communication at 12 months between the EUC (Arm A) and CONCURxP (Arm B) arms.

VI. To compare self-efficacy for managing symptoms at 12 months between the EUC (Arm A) and CONCURxP (Arm B) arms.

VII. To compare financial worry at 12 months between the EUC (Arm A) and CONCURxP (Arm B) arms.

EXPLORATORY OBJECTIVES:

I. To assess longitudinal changes of patient-reported outcomes (self reported adherence, symptom burden, quality of life, and financial worry) from the EUC (Arm A) and CONCURxP (Arm B) arms.

II. To compare healthcare utilization at 12 months between the EUC (Arm A) and CONCURxP (Arm B) arms.

III. To compare progression-free survival at 12 months between the EUC (Arm A) and CONCURxP (Arm B) arms.

IV. To compare overall survival at 12 months between the EUC (Arm A) and CONCURxP (Arm B) arms.

V. To describe CONCURxP (Arm B) patients and their provider experience with various implementation outcomes.

OUTLINE: Patients are randomized into 1 of 2 arms. Non-patient participants are assigned to arm C.

ARM A: Patients use the WiseBag medication dispenser and receive access to educational materials every 4 weeks over 12 months.

ARM B: Patients use the WiseBag medication dispenser and receive personalized text message reminders, medication tracking and healthcare provider follow ups as part of the CONCURxP platform over 12 months. Patients may complete an interview over 20-30 minutes within 6 months of study completion.

ARM C: Participants complete an interview over 20-30 minutes 15-39 months post-first patient enrollment.

After completion of study intervention, patients may be followed up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* NON-PATIENT: Participants must be an oncology healthcare provider (i.e., oncologist, advanced practice provider, or oncology nurse)
* NON-PATIENT: Participants must have taken care of at least one patient randomized to Arm B (CONCURxP) who had less than 85% adherence rate at 12 months as measured by the WiseBag
* NON-PATIENT: Participant must speak English
* NON-PATIENT: Participant must be employed at an National Cancer Institute Community Oncology Research Program (NCORP) site for at least 6 months
* NON-PATIENT: Participant must be able to provide informed consent to participate in this study
* PATIENT STEP 0: Patient must be >= 18 years of age
* PATIENT STEP 0: Patient must be fluent in written and spoken English OR patient must be fluent in written and spoken Spanish
* PATIENT STEP 0: Patient must present with new or established pathologically proven hormone receptor (HR)+ HER2- metastatic breast cancer at the time of Step 0
* PATIENT STEP 0: Patient must have initiated any of the CKD4/6 inhibitors (palbociclib or Ibrance, ribociclib or Kisqali, abemaciclib or Verzenio) within 30 days prior to consenting to Step 0 or have received a prescription order with stated intent to initiate within 30 days following Step 0 consent

  * NOTE: Patients who have been treated previously with anticancer treatments other than CDK4/6 inhibitors are eligible
  * NOTE: CDK4/6 inhibitors must be provided/supplied as a single agent blister pack. If the medication is supplied as capsules in a pill bottle (e.g., Ibrance capsules), patient is not eligible
  * NOTE: Ribociclib (Kisqali) and abemaciclib (Verzenio) are only available in blister packs. Palbociclib (Ibrance) is the only CDK4/6 inhibitor that might be available in a capsule formulation. However, this is an outdated formulation and is rarely prescribed as a new start. The format of ordered palbociclib can be determined based on the prescription order
* PATIENT STEP 0: Patients must not have been previously treated with any of the following CDK4/6 inhibitors: Palbociclib or Ibrance, ribociclib or Kisqali, and abemaciclib or Verzenio
* PATIENT STEP 0: Patients must not already be enrolled in a therapeutic clinical trial that monitors CDK4/6 inhibitors
* PATIENT STEP 0: Patient must confirm that they intend to receive their care or monitoring at an NCORP site
* PATIENT STEP 0: Patient must have a personal mobile phone in which they are able and willing to send and receive text messages

  * NOTE: The restriction to those with mobile phone access with text messaging is based on the primary intention of the study which involves the use of text messaging to improve adherence
* PATIENT STEP 0: Patient must have an email address

  * NOTE: The restriction to those with an email address is based on the primary intention of the study which involves patients responding to questions regarding their reasons for non-adherence after every missed dose to improve adherence
* PATIENT STEP 0: Patient must have the ability to understand and the willingness to sign a written informed consent document

  * NOTE: Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available are not eligible
* PATIENT STEP 0: Patient must not have an Eastern Cooperative Oncology Group (ECOG) performance status >= 3 OR patient must not be deemed medically unable to participate in the study by the study investigators or an oncology clinician (i.e., referral to hospice)
* PATIENT STEP 0: Patient must not be enrolled in other trials offering financial assistance

  * NOTE: Gift cards for survey completion, parking passes, or free medication provided as part of therapeutic trials are not considered financial assistance
* PATIENT STEP 1: Patient must meet all the eligibility criteria for Step 0
* PATIENT STEP 1: Patient must have signed a written informed consent form
* PATIENT STEP 1: Patient must have completed baseline survey within 30 days of the date of Step 0 Registration
* PATIENT STEP 1: Patients must have initiated their CDK 4/6 inhibitors within 30 days of the date of Step 0 registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Adherence using electronic monitoring | At 12 months after initiation of medication
  For each arm, mean and standard deviation (SD) adherence rates for all patients will be calculated. A two-sample t-test will be used to compare CDK4/6 inhibitor (CDK4/6i) adherence between the two arms at 12 months.

SECONDARY OUTCOMES:
Adherence using self-report | At 3, 6, and 12 months
  Using the12-item Patient Reported Outcomes Measurement Information System (PROMIS) Medication Adherence Scale compare mean score and changes in mean scores (from baseline) at each time point between the arms using two-sample t-tests.
CDK4/6i persistence | At 12 months after initiation of medication
  Defined as duration from CDK4/6i initiation to discontinuation of medication against medical advice, measured as the number of days from initiation until the first day of a gap that is 30 days or longer. For each arm, mean days of persistence, and the proportion of patients who discontinue the medication earlier than 12-month will be calculated and compared between the two arms using the two-sample t-test and chi-squared test, respectively.
Symptom burden | At baseline, 3, 6 and 12 months
  Using the 16-item National-Comprehensive Cancer Network Functional Assessment of Cancer Therapy Breast Cancer Symptom index compare mean score and changes in mean scores (from baseline) at each time point between the arms using two-sample t-tests.
Quality of life | At baseline and 12 months
  Using the PROMIS-10- version (v)1.2-Global Health compare mean score and changes in mean scores (from baseline) at each time point between the arms using two-sample t-tests.
Patient-provider communication | At baseline, 3, 6, and 12 months
  Using the Consumer Assessment of Healthcare Providers and Systems compare mean score and changes in mean scores (from baseline) at each time point between the arms using two-sample t-tests.
Self-efficacy for managing symptoms | At baseline, 3, 6, and12 months
  Using PROMIS Item Bank v1.0 - Self-Efficacy for Managing Symptoms compare mean score and changes in mean scores (from baseline) at each time point between the arms using two-sample t-tests.
Financial worry | At baseline, 3, 6, and12 months
  Using the Comprehensive Score for Financial Toxicity compare mean score and changes in mean scores (from baseline) at each time point between the arms using two-sample t-tests.

OTHER OUTCOMES:
Longitudinal changes of patient-reported outcomes | At baseline, 3, 6 and 12 months
  Generalized estimating equation will be used to assess the longitudinal change over time.
Healthcare utilization | At baseline, 3, 6, and12 months
  The difference of healthcare utilization between two arms will first be evaluated using the two sample t test for the continuous variables (e.g., length of stay or number of emergency department visits), and then be modeled through the regressions to allow for the control of other covariates if needed.
Progression-free survival | At 3 and 12 months
  Kaplan-Meier curves and log-rank testing will be used to visualize and compare progression free survival between the connected customized treatment platform (CONCURxP) patient group and enhanced usual care group, and Cox proportional hazards model will be fit to evaluate the impact of potential moderators on the associations of progression-free survival with arms.
Overall survival | At 3 and 12 months
  Kaplan-Meier curves and log-rank testing will be used to visualize and compare overall survival between the CONCURxP patient group and enhanced usual care group, and Cox proportional hazards model will be fit to evaluate the impact of potential moderators on the associations of overall survival with arms.
CONCURxP arm patients and their provider experience | Up to 12 months
  We will measure portal usability using patient-reported survey and will report mean and SD. For qualitative interviews, we will use conventional content analysis methods.
Characteristics of National Cancer Institute Community Oncology Research Program (NCORP) site patient population and the enrollees in EAQ221CD. | Up to 12 months
  Cox proportional hazards model will be fit to evaluate the impact of potential moderators (e.g., sociodemographic, insurance, cancer variables, endocrine therapy adherence, health literacy, health belief, medical history and NCORP practice characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Gelareh Sadigh, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (400):
- United States (393):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Mercy Cancer Center, Merced, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - BASS Medical Group - Lennon, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Mercy Health - Paducah Medical Oncology and Hematology, Paducah, Kentucky
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates, Baton Rouge, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Mississippi Baptist Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Hackettstown Medical Center, Hackettstown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Newton Medical Center, Newton, New Jersey
  - Chilton Medical Center, Pompton, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Westchester Emergency Center, Midlothian, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Bon Secours Richmond Community Hospital, Richmond, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Jefferson Healthcare, Port Townsend, Washington
  - Valley Medical Center, Renton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Ascension Saint Francis Hospital, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - Marshfield Medical Center - Neillsville, Neillsville, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Puerto Rico (7):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Sadigh G, Duan F, Gareen IF, Hancock J, Sicks JD, Thangarajah M, Meisel JL, Torres MA, Ramsey SD, Wolff AC, Wagner LI, Carlos RC, Graetz I. Improving CDK4/6 inhibitors adherence in breast cancer using the CONnected CUstomized Treatment Platform (CONCURxP) mobile health intervention: Study protocol for ECOG-ACRIN EAQ221CD. Contemp Clin Trials. 2026 Jan;160:108145. doi: 10.1016/j.cct.2025.108145. Epub 2025 Nov 18. PMID 41265834